CLINICAL TRIAL: NCT01138592
Title: Pilot Study to Evaluate the Clinical Utility of 3M Littmann Scope-to-Scope Software for Real-time Assessment of Patients at Remote Clinic Locations by Centrally-located Medical Providers
Brief Title: Pilot Study to Evaluate the Clinical Utility of Auscultation Software at Remote Locations
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-003041
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Auscultation of Heart and Lungs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Care Patients: Any patient undergoing a telemedicine evaluation involving auscultation of the heart and lungs.

SUMMARY:
Primary Objective: Evaluation of the utility of real-time, scope-to-scope communication between commercially-available 3M Littmann Electronic Model 3200 Electronic stethoscopes over a dedicated intranet system for the assessment of patients at remote (satellite) clinic locations by centrally-located (hub) medical providers.

Secondary Objective: Comparison of the accuracy of patient assessment between the remotely located, mid-level presenter with the centrally-located physician or nurse practitioner provider.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects who are at least 18 years of age
2. Subjects who are scheduled to undergo examination in a telemedicine setting
3. Subjects who are willing to voluntarily sign the compound Informed Consent and the Authorization to Disclose Protected Health Information Form.

Exclusion Criteria:

1. Subjects who are unwilling to undergo additional examination in a telemedicine setting,
2. Any subject requiring time-critical medical intervention.
3. Any subject who the investigator believes should not be included or is unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Patients Hepatitis C Patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Confirmation of hub (remote) observations with satellite (local) observations | 30 minutes
  Presence or absence of heart or lung sound; e.g., murmurs, etc., and/or rales, rhonchii, wheezes.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Henley, MD, MPH, Principal Investigator — North Country Health Care, Flagstaff, AZ
Locations (1):
- North Country Health Care, Flagstaff, Arizona, United States